



## **Consent Form**

| Project Title | An exploratory study on the prevalence of sarcopenia- |
|---|---|
| | promoting medicines in people with sarcopenia and falls |
| Principle investigator name | Kamaldeep Sahota |
| Patient Identification for project | |

| | | Please<br>initial |
|---|---|---|
| 1. | I confirm that I have read and understood the information sheet dated July 2025 (Version 4) for the above study and have had the opportunity to ask questions | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from (company name) or from regulatory authorities, or NHS Trust where it is relevant to my taking part in the research. I permit these individuals to have access to my records. | |
| 4. | I agree to take part in the above study. | |
| 5. | Optional: I would like to receive a summary of the results when the study is finished. [Yes / No] (please circle). If yes, please provide your preferred contact details: | |

| Name of participant |
|---------------------|
| Date |
| Signature |





| Name of person taking consent |
|-------------------------------|
| Date |
| Signature |

Please complete in duplicate and allocate 1 form for the Patient and 1 to be kept as part of the study documentation.